CLINICAL TRIAL: NCT07252869
Title: Evaluation of the Accuracy of Intraoral Scanner Versus Analog Impression in Implant Supported Rehabilitations Performed With Flapless Computer-Guided Implantology
Brief Title: Evaluation of Impression Accuracy: Digital Scanner Versus Analog Technique
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Stefano Storelli, Reasearcher, University of Milan
Other Study IDs: 1361
Record Dates: First submitted 2025-05-21; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-05

CONDITIONS: Accuracy and Precision of Noninvasive Measurement
MeSH Terms: interventions — Inosine Monophosphate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TRIOS®-3Shape Group: Participants whose models were scanned using the TRIOS®-3Shape intraoral digital scanner. The deviation from the reference model was calculated to assess the accuracy of this technique.
  Interventions: Other: Digital impression
- CS 3600® Carestream Group: Participants whose models were scanned using the CS 3600® Carestream Dental intraoral scanner. The deviation from the reference model was analyzed to evaluate the technique's precision.
  Interventions: Other: Digital impression
- PVS Analog Impression Group: Participants whose impressions were taken using conventional polyvinylsiloxane (PVS) material. Cast models were scanned and compared to the reference to determine the accuracy of analog impressions.
  Interventions: Other: impression

INTERVENTIONS:
Other: impression — A Comparative Study of Digital Versus Analog Impressions
  Groups: PVS Analog Impression Group
Other: Digital impression — impression taken by intraoral scanner
  Groups: CS 3600® Carestream Group; TRIOS®-3Shape Group

SUMMARY:
The goal of this study is to evaluate the accuracy of intraoral impressions obtained using the Trios 3Shape® and Carestream CS 3600™ scanners, as well as traditional analog impressions using polyvinyl siloxane (PVS), in comparison to a gold standard represented by a laboratory scanner in 51 dental models from 42 patients affected by partial edentulism who required at least two implants.

Researchers compare Trios 3Shape®, Carestream CS 3600™ and polyvinyl siloxane (PVS) to see if there is a different accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* Implant placement in healed bone sites (at least 8 weeks post-tooth extraction or at least 6 months after regenerative procedures), allowing guided implant insertion of at least 3.3 mm in diameter or 8.5 mm in length;
* Implant site without ongoing infections or dental extraction residues;
* Good systemic health conditions and adequate oral hygiene;
* Periapical and periodontal health of opposing teeth/implants in occlusion;
* Edentulism of at least two adjacent dental elements.

Exclusion Criteria:

* Ongoing diseases requiring prolonged use of corticosteroids;
* Leukocyte dysfunction or deficiencies;
* Severe hemophilia;
* Current pregnancy;
* Past and/or current head/neck radiotherapy and/or chemotherapy;
* Renal insufficiency;
* Past and/or current use of bisphosphonates;
* Uncompensated endocrine disorders;
* Physical disabilities preventing adequate oral hygiene;
* Alcohol abuse and drug use;
* Smokers (>10 cigarettes/day);
* Untreated periodontitis;
* Mucosal diseases (e.g., erosive Lichen Planus);
* Severe parafunctional habits (e.g., bruxism or clenching);
* Persistent intraoral infections;
* Allergies or adverse reactions to restorative materials;
* Completely edentulous arches;
* Limited mouth opening;
* Inadequate oral hygiene or lack of motivation for self-care;
* Uncontrolled systemic diseases;
* Untreated or chronic oral cavity diseases;
* Fully edentulous arches.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients seeking implant treatment at the Implantology and Prosthodontics Department of the Giorgio Vogel Odontostomatological Clinic, ASST Santi Paolo e Carlo, Milan.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical and radiological evaluation of soft tissues and bone level in implant supported rehabilitations performed with Flapless Computer-Guided implantology. A prospective clinical study. | Patients included in this prospective study were recruited from 2017 to 2022
  The statistical analyses were performed using AnalystSoft StatPlus®. Using GOM Inspect by Zeiss®, the mean deviation values from the reference file were calculated for each model. They were expressed in absolute terms. In our study, for each of the three test techniques (TRIOS®-3Shape, CS 3600® Carestream Dental, and PVS), the average of the values obtained from the superimpositions of 51 models was calculated, resulting in the mean deviation of each method from the reference.
  For data analysis, a one-way ANOVA test and a two-sample Z-test were applied, with a significance level (α) set at 0.05. These tests were used both to compare the mean distances and to assess the standard deviations of the deviations. Each technique was considered accurate if its mean deviation was less than 30 μm.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontoiatrica Giorgio Vogel (Università degli studi di Milano), Milan, Italy, Italy